CLINICAL TRIAL: NCT06786871
Title: ARTLifeLine: Assisted Reproduction Technology (ART) Family Health and Development Trajectory Cohort (ARTLL)
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023095
Record Dates: First submitted 2023-06-20; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-06

CONDITIONS: Reproductive Techniques, Assisted; Family; Cohort Studies; Development, Infant; Reproductive Issues
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Couples who have had or plan IVF fertility treatment and their offsprings: Have performed or plan to undergo IVF fertility treatment; Paper or electronic medical records during fertility treatment are available; Obtain informed consent from the research subject or guardian of the minor
  Interventions: Procedure: IVF treatment

INTERVENTIONS:
Procedure: IVF treatment — Methods or procedures for the in vitro processing of human oocytes, sperm, or embryos for fertility purposes

SUMMARY:
The goal of this observational study is to study the health status of infertile couples and their offspring using assisted reproductive technologies. The main questions it aims to answer are:

1. On the basis of the assisted reproduction birth cohort and related research established by the team in the early stage, further expand the construction of the "tracking cohort of familial health and development using assisted reproduction", combine emerging technologies such as cross-database linking and integration, multi-omics sequencing and classical cohort research design, and carry out long-term longitudinal follow-up across generations, covering the whole life cycle and health in multi-dimension.
2. Build a disease risk prediction model for pregnant women and children with assisted reproduction.
3. Delineate the growth curve and neurobehavioral development trajectory of assisted reproductive offspring at different stages.
4. Evaluate the adolescent fertility potential and risk factors of assisted reproductive offspring.

DETAILED DESCRIPTION:
1. Recent Research Objectives (Within Five Years):

   Build a risk prediction model for reproductive women and children in assisted reproduction, and identify potential molecular markers with high predictive value to provide epidemiological evidence clues for further basic mechanism research.

   Analyze the health status of natural conception versus assisted reproduction pregnant women and children, growth and developmental curves of fetuses during pregnancy, and early neurobehavioral development levels of children after birth.
2. Medium to Long-Term Research Objectives (Future Research Directions of the Cohort):

Systematically evaluate the long-term effects of infertility and assisted reproductive treatments on the physiological, psychological, individual, and family development of parents and offspring.

Collaborate and share data with other domestic and international health cohorts or databases related to assisted reproduction, to compare and analyze the long-term safety of various assisted reproductive technologies on the health of infertile couples and their offspring.

ELIGIBILITY:
Inclusion Criteria:

(1) Previous or planned IVF treatment; (2) paper or electronic medical records during fertility treatment are available; (3) Obtain informed consent from the research subject or guardian of the minor.

Exclusion Criteria:

(1) Other assisted reproductive treatment techniques that exclude in vitro fertilization, including guided intercourse, ovulation induction, artificial insemination, etc.; (2) refusal of enrollment; (3) withdraw or abort the study at any time and for any reason.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Couples who have had or plan IVF fertility treatment and their children. Study is recruitign on a family-by-family basis, including: couples undergoing IVF for a variety of reasons, children born as a result of IVF treatment, and other children in the family
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Health outcomes | 20 years
  Health outcomes for parents and children at different stages(assisted reproduction Treatment stage, pregnancy and childbirth, childhood, adolescence) and dimensions(physiological, psychological, individual and family development) after receiving assisted reproduction treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, PhD, Study Chair — Peking University Third Hospital; Rong Li, PhD, Study Director — Peking University Third Hospital; Wei Yuan, PhD, Principal Investigator — Peking University Third Hospital; Tongyan Han, PhD, Principal Investigator — Peking University Third Hospital; Liying Yan, PhD, Study Director — Peking University Third Hospital; Yuanyuan Wang, PhD, Principal Investigator — Peking University Third Hospital; Rui / Yang, PhD, Principal Investigator — Peking University Third Hospital; Xiaohui / Zhu, PhD, Principal Investigator — Peking University Third Hospital; Lian / Chen, PhD, Principal Investigator — Peking University Third Hospital; Meihua / Piao, PhD, Principal Investigator — Peking University Third Hospital; Yunpu / Cui, PhD, Principal Investigator — Peking University Third Hospital; Yanan / Tang, PhD, Principal Investigator — Peking University Third Hospital; Chunling / Huang, PhD, Principal Investigator — Peking University Third Hospital; Chunmei / Zhang, PhD, Principal Investigator — Peking University Third Hospital; Linlin / Wang, PhD, Principal Investigator — Peking University Third Hospital; Ningning / Pan, PhD, Principal Investigator — Peking University Third Hospital; Huifeng Shi, PhD, Principal Investigator — Peking University Third Hospital; Tianchen / Wu, PhD, Principal Investigator — Peking University Third Hospital; Wanning / Qiu, PhD, Principal Investigator — Peking University Third Hospital; Jinfang / Yuan, PhD, Principal Investigator — Peking University Third Hospital; Hui / Zhang, MD, Principal Investigator — Peking University Third Hospital; Qingqing Wang, Principal Investigator — Peking University Third Hospital; Meng Qin, Principal Investigator — Peking University Third Hospital; Ying Kuo, Principal Investigator — Peking University Third Hospital; Wenxi Zhang, Principal Investigator — Peking University Third Hospital; Shuo Guan, Principal Investigator — Peking University Third Hospital; Siming Jiang, Principal Investigator — Peking University Third Hospital; Fei Kong, Principal Investigator — Peking University Third Hospital; Tian Tian, PhD, Principal Investigator — Peking University Third Hospital; Lixue Chen, Principal Investigator — Peking University Third Hospital; Yu Fu, Principal Investigator — Peking University Third Hospital; Fang Liu, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, China, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No